CLINICAL TRIAL: NCT00825604
Title: Quality of Life and Achievement of Target of Treatment After Optimized Medical Treatment, Physical Training and Smoking Cessation With or Without Percutaneous Coronary Intervention in Patients With Stable Angina Pectoris.
Brief Title: Quality of Life and Target Achievement After Treatment of Patients With Stable Angina Pectoris
Acronym: LOBSTR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of poor inclusion difficulties to find patient
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr: 056-08
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Stable Angina Pectoris
Keywords: stable coronary artery disease; quality of life; target achievement; physical training; percutaneous coronary intervention
MeSH Terms: conditions — Angina, Stable | interventions — Angioplasty, Balloon, Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without PCI (No Intervention): Optimized medical treatment, physical training and smoking cessation
- With PCI (Active Comparator): optimized medical treatment, physical training and smoking cessation with complimentary treatment with percutaneous coronary intervention(PCI)
  Interventions: Procedure: Percutaneous coronary angioplasty (PCI)

INTERVENTIONS:
Procedure: Percutaneous coronary angioplasty (PCI) — optimized medical treatment, physical training and smoking cessation with complimentary treatment with coronary angioplasty (PCI):
  Other Names: PCI
  Arms: With PCI

SUMMARY:
The purpose of this study is to, in patients with stable angina pectoris, assess the additional benefit of PCI on top of optimized medical treatment, physical training and smoking cessation with regard to quality of life, achievement of target of treatment and clinical events such as death, acute myocardial infarction, stroke and revascularization.

DETAILED DESCRIPTION:
Patients with stable angina pectoris with a significant coronary stenosis will be randomized to optimized medical treatment, physical training and smoking cessation or to optimized medical treatment, physical training, smoking cessation and complimentary treatment with PCI. All patients will be followed up at six months and at one and five years regarding symptoms, blood lipids, systemic blood pressure, physical training status, smoking habits, and maximal exercise ECG.

Achievement of target of treatment will be measured by questions regarding the patients' expectation of the treatment at baseline and at a 6 month follow-up. The questions at 6 months will be based on the interviews at inclusion. Furthermore quality of life will be measured with three different measuring instrument; SF-36 short form, Seattle Angina Questionnaire (SAQ), and EQ-5D. These instruments will be given to the patients at baseline, at six months and at the five year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease
* Angina pectoris with at least angina class 2 according to Canadian Cardiovascular Society (CCS)
* Angiographic verified stenos in a native vessel
* Accepted for PCI

Exclusion Criteria:

* Instable coronary artery disease or AMI withín two months
* CCS class IV
* Stenosis in Left main and/or proximal LAD
* NYHA- III-IV
* Fall in blood pressure during exercise test > 10mm Hg, measured two times
* Contraindication or allergy against clopidogrel or ASA
* Unable to communicate verbal or i writing
* Unwillingness to participate in the study
* Participating in an other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Quality of life measured by SF36 | 6 months

SECONDARY OUTCOMES:
Achievement of target of treatment based on interview of the patients | 6 months
Death, myocardial infarction, stroke or new revascularization | 6 months, one year and five years after randomization
To assess expectations of treatment at inclusion and fulfilment of expectations | 6 months
Quality of life measured by EQ5D and Seattle angina questionaire | 6 months and 5 years
Health economy | 6 months, one year and five years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grip, Prof., Principal Investigator — Göteborgs Universty
Locations (1):
- Sahlgrenska University hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127
- [Background] Henderson RA, Pocock SJ, Clayton TC, Knight R, Fox KA, Julian DG, Chamberlain DA; Second Randomized Intervention Treatment of Angina (RITA-2) Trial Participants. Seven-year outcome in the RITA-2 trial: coronary angioplasty versus medical therapy. J Am Coll Cardiol. 2003 Oct 1;42(7):1161-70. doi: 10.1016/s0735-1097(03)00951-3. PMID 14522473
- [Background] Pitt B, Waters D, Brown WV, van Boven AJ, Schwartz L, Title LM, Eisenberg D, Shurzinske L, McCormick LS. Aggressive lipid-lowering therapy compared with angioplasty in stable coronary artery disease. Atorvastatin versus Revascularization Treatment Investigators. N Engl J Med. 1999 Jul 8;341(2):70-6. doi: 10.1056/NEJM199907083410202. PMID 10395630
- [Background] Weintraub WS, Spertus JA, Kolm P, Maron DJ, Zhang Z, Jurkovitz C, Zhang W, Hartigan PM, Lewis C, Veledar E, Bowen J, Dunbar SB, Deaton C, Kaufman S, O'Rourke RA, Goeree R, Barnett PG, Teo KK, Boden WE; COURAGE Trial Research Group; Mancini GB. Effect of PCI on quality of life in patients with stable coronary disease. N Engl J Med. 2008 Aug 14;359(7):677-87. doi: 10.1056/NEJMoa072771. PMID 18703470
- [Background] Sullivan M, Karlsson J. The Swedish SF-36 Health Survey III. Evaluation of criterion-based validity: results from normative population. J Clin Epidemiol. 1998 Nov;51(11):1105-13. doi: 10.1016/s0895-4356(98)00102-4. PMID 9817128
- [Background] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Fihn SD. Monitoring the quality of life in patients with coronary artery disease. Am J Cardiol. 1994 Dec 15;74(12):1240-4. doi: 10.1016/0002-9149(94)90555-x. PMID 7977097
- [Background] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, Fihn SD. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995 Feb;25(2):333-41. doi: 10.1016/0735-1097(94)00397-9. PMID 7829785
- [Background] Sullivan M, Karlsson J, Ware JE Jr. The Swedish SF-36 Health Survey--I. Evaluation of data quality, scaling assumptions, reliability and construct validity across general populations in Sweden. Soc Sci Med. 1995 Nov;41(10):1349-58. doi: 10.1016/0277-9536(95)00125-q. PMID 8560302
- [Background] Jones B, Jarvis P, Lewis JA, Ebbutt AF. Trials to assess equivalence: the importance of rigorous methods. BMJ. 1996 Jul 6;313(7048):36-9. doi: 10.1136/bmj.313.7048.36. PMID 8664772
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Hambrecht R, Walther C, Mobius-Winkler S, Gielen S, Linke A, Conradi K, Erbs S, Kluge R, Kendziorra K, Sabri O, Sick P, Schuler G. Percutaneous coronary angioplasty compared with exercise training in patients with stable coronary artery disease: a randomized trial. Circulation. 2004 Mar 23;109(11):1371-8. doi: 10.1161/01.CIR.0000121360.31954.1F. Epub 2004 Mar 8. PMID 15007010